CLINICAL TRIAL: NCT03086733
Title: Phase II Study of Single Agent Pre-operative Metformin in Patients With Clinical Stage I - IIIA NSCLC Proceeding to Surgical Resection. 'Lung Metcore Study'
Brief Title: Phase II Lung Metcore - Preoperative Metformin for Lung Cancer
Acronym: Metcore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-9560.0 - Lung Metcore Study
Record Dates: First submitted 2017-02-24; First posted 2017-03-22 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Lung Cancer; Non small cell lung cancer; Metformin; Pre-operative treatment; Neoadjuvant treatments; Cancer; Phase II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: single center, open label, single arm Phase II study of a pre-operative window of metformin treatment in stages I - IIIA NSCLC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Metformin (Experimental): 14 to 21 days of pre-operative Metformin tablets First 5 days 850 mg OD v/o 850 mg BID thereafter until 21 days are completed.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg tablets v/o OD for first 5 days 850 mg tablets v/o BID until day 21
  Other Names: Glucophage

SUMMARY:
This is a phase II single centre open label single arm pre-operative window of metformin treatment in stage I-IIIa Non small cell lung cancer.

In which patients will be invited to participate by receiving Metformin treatment during 14 to 21 days at 850 mg BID until the day before surgery.

They will be followed closely for any Adverse Events during treatment and 30 days after surgery. During treatment there will be no follow up tests except 1 fasting blood glucose at week 2 of treatment.

Survival data will be prospectively gathered after study treatment has ended until death.

DETAILED DESCRIPTION:
Title of study: Phase II study of single agent pre-operative metformin in patients with clinical stage I - IIIA NSCLC proceeding to surgical resection. 'Lung Metcore Study'

Objectives:

To evaluate the effects of short-term pre-operative exposure to metformin in operable stages I to IIIA NSCLC.

Primary end-points:

* The difference in the proportion of proliferating NSCLC cells (measured by comparing Ki67 levels) prior to and after metformin treatment.
* The rate of apoptosis of NSCLC (measured by the TUNEL assay) prior to and after metformin treatment.

Secondary end-points:

* The safety and tolerability of preoperative metformin administration in NSCLC, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE [version 4.0])
* Pathologic changes in lung tissue after metformin administration. Study Design: This trial is designed as a single center, open label, single arm Phase II study of a pre-operative window of metformin treatment in stages I - IIIA NSCLC. The efficacy of metformin will be assessed by its effects on markers of cellular proliferation and apoptosis. Exploratory analysis of molecular markers of the hypothesized effects of metformin in NSCLC will also be carried out. Furthermore, changes in serum ligands to growth signaling pathways in lung cancer with metformin treatment will be measured.

Number of patients: Thus, the total expected sample size is approximately 50 patients, anticipating minimal loss of eligible participants through treatment intolerance or acceleration of surgery. Accrual is estimated at 1.5 to 2 patients per month for 25 to 33 months, based on accrual rates for a recent pre-operative window thoracic surgical study at UHN.

• Metformin will be started at a dose of 850mg daily then increased to 850mg b.i.d. (morning and evening) after 5 days as tolerated. Treatment will be given from the time of enrollment till the evening prior to surgery.

Correlatives:

The following molecular and serological correlative biomarkers will be considered covariates in the analysis of primary endpoints of the phase II study. Covariate pretreatment values and changes in covariate values (where applicable) will be used to estimate the relationship between covariates and patient's Ki67 or apoptotic response using logistic regression. It is noted that several covariates are being tested and the number of patients being analyzed is small, thus, some tests may be statistically significant due to chance even if no association exists.

* Genetic Mutations in NSCLC (On pre-treatment biopsies by molecular techniques):

  * LKB1 mutational status (Sequencing)
  * EGFR, Ras, AKT, PI3K mutations (Oncocarta platform)
  * EGFR gene copy number (FISH)
  * ALK rearrangement status
* Protein Marker of Resistance To Metformin (On pre-treatment biopsies by immunohistochemistry

  * OCT1 expression
  * PROTEIN MARKERS OF RECEPTORS AND ACTIVATED PATHWAYS TO mtor IN NSCLC (Comparison between pre-treatment biopsies and post-resection specimens by immunohistochemistry):
  * IR
  * IGF-1R
  * Phosphorylated-AMPK
  * EGFR and phospho-EGFR
  * PKB (AKT) and phospho-AKT
  * Phosphorylated (erbb2, erbb3, erbb4)
  * Phosphorylated-STAT3
  * Phospho-ribosomal protein S6
* VASCULARITY IN NSCLC (Comparison between pre-treatment biopsies and post-resection specimens by immunohistochemistry):

  * VEGF
  * Microvessel density count (CD34, CD105)
* SERUM LIGANDS TO SIGNALLING PATHWAYS IN NSCLC (Comparison between pre-treatment biopsies and post-resection specimens by ELISA):

  * Insulin
  * Glucose
  * IGF-1
  * TGF-α
  * TNF-α
  * Calculated HOMA
  * CRP
  * Adiponectin

Statistics:

Patients who completed metformin treatment will have the Ki67 and apoptosis scores compared between samples obtained pre and post-metformin treatment. Changes in Ki67 and apoptotic scores with metformin treatment will be correlated with the biomarkers of various pathways hypothesized to mediate an effect of metformin on NSCLC development.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy-proven non-small cell lung carcinoma (NSCLC) of any histological variant except for neuroendocrine tumors. Patients must not have mixed NSCLC and small cell lung cancer (SCLC).
* Be of clinical stage I to IIIA (according to the 7th lung cancer TNM classification and staging system) by radiologic and/or pathologic criteria where appropriate (e.g. mediastinoscopic staging). Baseline CT-chest scan must be within 4 weeks of study entry.
* Be deemed appropriate candidates for surgical resection by the treating surgeon and assessing team.
* Be aged - 18 years or more.
* Have ECOG performance status - 2.
* Have organ and marrow function as defined below for safe lung biopsy and administration of metformin:

  * Platelets -100 000
  * Total bilirubin -1.5 X institutional upper limit of normal
  * AST/ALT -2 X institutional upper limit of normal
  * Creatinine clearance -60 mL/min/1.73 m2
* Have the ability to understand and the willingness to sign a written informed consent document.
* Not require emergency surgery within 14 days of staging investigations.
* Not have received anticancer treatment with chemotherapy, radiotherapy or Epidermal - - Growth Factor Receptor (EGFR) inhibitor therapy for the current lung cancer.
* Not have a concomitant active malignancy or be receiving any other investigational or anticancer agents while on the study, to avoid the influence of alternative anti-cancer therapy. Otherwise, those with a past history of cancer are eligible.

Exclusion Criteria:

* Not have a past history of an allergic reaction to metformin.
* Not have a past history of diabetes mellitus or fasting glucose ≥ 7.0 mmol/L.
* Not have a past history of lactic acidosis or metabolic acidosis.
* Not have consumption of ≥ 3 alcoholic beverages per day (average).
* Not have had regular use of agents that may influence insulin sensitivity/levels within 4 weeks of study entry.
* Not have uncontrolled intercurrent illness (es) including but not limited to: ongoing or active:

  * Infection,
  * Symptomatic congestive
  * Cardiac failure or evidence of cardiac dysfunction,
  * Unstable angina pectoris,
  * Cardiac arrhythmia,
  * Active peptic ulcer disease or gastrointestinal conditions (e.g. Inflammatory bowel disease) or
  * Psychiatric illness/social situations that would limit compliance with study requirements.
* Not be on a loop diuretic due to their potential to cause renal impairment and predispose to lactic acidosis.
* Not have contrast-enhanced imaging (except when clinically indicated) while on the study. Iodinated contrast agents can cause renal failure, leading to metformin accumulation and lactic acidosis.
* Women should not be pregnant or become pregnant during study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Ki67 | 45 days after surgery
  • The difference in the proportion of proliferating NSCLC cells (measured by comparing Ki67 levels) prior to and after metformin treatment.
Apoptosis | 45 days after surgery
  • The rate of apoptosis of NSCLC (measured by the TUNEL assay) prior to and after metformin treatment.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | During a minimum of 14 days and maximum of 21 days patients will be assessed every 5 days during treatment and 30 days after surgery
  • The safety and tolerability of preoperative metformin administration in NSCLC, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE [version 4.0])
Pathology | 45 days after surgery
  • Pathologic changes in lung tissue after metformin administration

CONTACTS AND LOCATIONS:
Overall Officials: Tom Waddell, MD, Principal Investigator — Head of Thoracic Surgery Division
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided